CLINICAL TRIAL: NCT01494519
Title: A Prospective Randomized Trial to Assess Fixation Strategies for Severe Open Tibia Fractures:Modern Ring External Fixators Versus Internal Fixation
Brief Title: Assessment of Fixation Strategies for Severe Open Tibia Fractures
Acronym: FIXIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-09-2-0108
Record Dates: First submitted 2011-08-25; First posted 2011-12-19 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Severe Open Fractures of the Tibia (Shin) Bone
Keywords: External ring fixation; internal fixation; traumatic tibia fracture
MeSH Terms: interventions — Surgical Procedures, Operative; Bone Plates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treament Arm 1 (Active Comparator): Definitive fixation with an external ring fixator.
  Interventions: Procedure: Surgery with an external ring fixator
- Treatment arm 2 (Active Comparator): Definitive fixation with a locked IM nail or plate
  Interventions: Procedure: Definitive fixation with a locked IM nail or plate

INTERVENTIONS:
Procedure: Surgery with an external ring fixator — Modern ring external fixator is defined as any fixator that has at least 1 ring proximal and 1 ring distal to the fracture site. The rings may be connected to the tibia using any combination of external fixation pins or wires at the surgeon's discretion. There must be at least two pins or wires connected to each ring, and typically there will be at least three pins or wires. Any FDA approved ring fixator meeting this definition from any manufacturer is allowed.
  Arms: Treament Arm 1
Procedure: Definitive fixation with a locked IM nail or plate — Eligible patients with tibial diaphyseal fractures will typically receive a standard locked IM Nail. The nail must use at least one static interlock proximal to and one static interlock distal to the fracture site. The nail may be placed with either a reamed or unreamed technique.
  Methaphyseal fractures, especially those with fracture lines extending into the joint may be more commonly treated with plate fixation. The plate may be applied in an open or percutaneous fashion. Any combination of locked and/or non-locked screws may be used.
  Arms: Treatment arm 2

SUMMARY:
The purpose of this study is to compare the use of modern ring external fixation versus internal fixation for fracture stabilization of severe open tibia fractures.

DETAILED DESCRIPTION:
Severe open fractures of the tibia (shin) bone are difficult to treat and are associated with high rates of infection and other complications. There is controversy regarding the best treatment, particularly in fractures with large wounds from trauma. The two current standard treatment options are to place an internal fixation device (a nail or plates with screws) or to use a device with pins that stick out of the skin and attach to rings outside the body (modern ring external fixator). It is unknown which of these standard of care treatment options will result in lower complication rates and better function of the leg.

Our goal is to perform a multi-center randomized controlled trial of the use of modern ring external fixation versus internal fixation for fracture stabilization of severe open tibia fractures. Patients who refuse randomization have the option of participating in a prospective observational study and the treatment is decided by the surgeon and patient.

Primary Aim: To compare the outcomes associated with modern ring external fixators versus standard internal fixation techniques in treating "severe" open tibia shaft or metaphyseal fractures with or without a bone defect of any size.

Primary Hypothesis: Among patients with open tibia shaft or metaphyseal fractures (with or without a bone defect of any size), the rate of re-hospitalization for major limb complications will be lower for patients treated with ring fixators than those treated with standard internal fixation.

Secondary Hypotheses: Among patients with open tibia shaft or metaphyseal fractures (with or without a bone defect of any size), the overall rate of infections will be lower for patients treated with ring fixators than those treated with standard internal fixation. Measures of fracture healing, limb function, and patient reported outcomes (including pain) will be as good or better among patients treated with ring fixators than those treated with standard internal fixation.

Secondary Aim #1: To determine the percentage of Gustilo IIIB open tibia shaft fractures that can be treated successfully (i.e. without amputation) without a soft tissue flap secondary to the use of ring external fixators.

Secondary Aim #2: To determine the two-year treatment costs associated with fixation of "severe" open tibia shaft or metaphyseal fractures (with or without a bone defect of any size) using modern ring external fixators versus standard internal fixation techniques.

Secondary Aim #3: To determine patient reported levels of satisfaction with the fixation method and overall treatment and to compare satisfaction between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. All open tibia fractures meeting at least one of 1 the following criteria:

   * Diaphyseal or metaphyseal Type IIIB (Gustilo IIIB Fractures are open fractures that require either a rotational or free flap for coverage of a soft tissue defect).
   * Diaphyseal or metaphyseal Type IIIA where extensive contamination or muscle damage (e.g. all military injuries from IED) precludes nail/plate placement at first debridement.
   * Diaphyseal or metaphyseal Type IIIA, where injury would have been classified as a IIIB, but because enough muscle was removed, the skin could be closed.
   * Diaphyseal or metaphyseal Type IIIA, where after debridement, bone gap is greater than 1cm.
   * Diaphyseal or metaphyseal Type IIIA, where fasciotomies were performed for impending or diagnosed compartment syndrome, and wounds could not be closed primarily (i.e. needs skin grafting).
2. Ages 18 - 64 years inclusive
3. Study fracture is suitable for limb salvage using either a modern ring external fixator or internal fixation (internal fixation =locked intramedullary nail or plate).

Inclusion notes:

1. Patients may have co-existing non-tibial infection, with or without antibiotic treatment.
2. Patients may have risk factors for infection including diabetes, immunosuppression from steroids or other medications, HIV, or other infections.
3. Patients may have a traumatic brain injury.
4. Patients may be treated initially with a temporary external fixator prior to randomization.
5. Patients may be treated initially at an outside institution prior to transfer to the study institution, as long as the definitive fixation was not performed prior to entrance into the study.
6. Patients with bilateral injuries that meet inclusion criteria may be included, but only the limb rated as "more severe" by the treating surgeon will be enrolled in the study.
7. Fractures may have a gap after debridement of any size, including no gap.

Exclusion Criteria:

1. Patients presenting with a traumatic amputation of the tibia
2. Patients already received definitive fixation with an IM nail, plate or ring fixator prior to study enrollment
3. Tibia already infected as diagnosed by a surgeon and currently receiving treatment for it
4. Patient speaks neither English nor Spanish
5. Patient is a prisoner
6. Patient has been diagnosed with a severe psychiatric condition
7. Patient is intellectually challenged without adequate family support
8. Patient lives outside the catchment area
9. Non-ambulatory patient due to an associated complete spinal cord injury
10. Non-ambulatory before the injury due to a pre-existing condition.
11. Complex pilon and plateau fractures. The study tibia fracture may have extension into the joint surface, but should primarily be a metaphyseal or diaphyseal fracture and not have an ipsilateral tibial plateau or pilon fracture.Contralateral tibial plateau and pilon fractures are allowed

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 442 (Actual)
Dates: Start 2011-07; Primary Completion 2017-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Re-hospitalization for Complication. | 2 years
  A hospital re-admission for a complication is defined as any re-admission to the hospital secondary to the treatment of the open tibia fracture for a defined set of complications. The list of complications includes: amputation (at any level), infection (defined using CDC criteria), flap failure, non-union, mal-union, loss of reduction, or hardware failure.

SECONDARY OUTCOMES:
Infection. | 2 years
  Infection is defined as either deep or superficial. The presence of tibia infection will be defined by the criteria of CDC. Deep infections are further defined as those that require operative treatment. Superficial infections are defined as those that are treated only with local antibiotics and wound care, and no operative treatment for the infection.
Fracture Healing. | 2 years
  Fractures will be evaluated with standard 2 view radiographs of the tibia as is currently performed in standard practice at every clinic visit after the 2 week follow-up. Fracture healing is measured by the treating surgeon using standard clinical criteria.
Limb Function. | 2 years
  Limb function will be measured using standard clinical assessments to include weight bearing and ambulation status, knee and ankle range of motion and self selected walking speed.
Patient Reported Outcome and Quality of Life. | 2 years
  Outcomes from the patients' perspective will be assessed using standardized questionnaires including the VR-12, the SMFA, and the Paffenbarger activity scale. Depression will be assessed using the PHQ. Post traumatic stress will be measured using the PCL-S.
Pain | 2 years
  Pain will be measured using the visual analogue scale (VAS), the brief pain inventory (BPI) and documentation of use of pain medications.
Satisfaction with treatment | 2 years
  Patient satisfaction with treatment will be measured using the Short Form Patient Satisfaction Questionnaire (PSQ-18).
Health Care Costs | 2 years
  Costs for the initial hospitalization and subsequent care will be estimated using electronic billing records and self reported health service utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Reider, MHS, PhD, Study Director — Major Extremity Trauma Research Consortium
Locations (33):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Naval Medical Center San Diego, San Diego, California
  - UCSF Medical Center, San Francisco, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - University of Miami Ryder Trauma Center, Miami, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Florida Orthopaedic Institute, Tampa General Hospital, Tampa, Florida
  - Eskenazi Health, Indianapolis, Indiana
  - OrthoIndy / Methodist Hospital, Indianapolis, Indiana
  - St Vincent Hospital, Indianapolis, Indiana
  - University of Maryland, R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Hennepin County Medical Center / Minneapolis, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Louis Medical Center, St Louis, Missouri
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Geisinger Health System, Danville, Pennsylvania
  - Penn State University M.S. Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - UT Health: The University of Texas Health Science Center at Houston Medical School, Houston, Texas
  - University of Texas Health Science Center, San Antonio, San Antonio, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - University of Wisconsin, Madison, Wisconsin